CLINICAL TRIAL: NCT06567288
Title: Effeect of Spencer Muscle Energy Technique on Pain in Diabetic Stiff Shoulder
Brief Title: Effect of Spencer Muscle Energy Technique on Pain in Diabetic Stiff Shoulder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed El-Moatasem Mohamed, lecturer of physical therapy, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004908
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- spencer muscle energy technique (Experimental): Spencer muscle energy technique (SMET) attempts to re-establish functional relationship between soft and articular tissues of the shoulder region, minimizes inflammatory and later developing fibrotic process, and restores arterial, venous, and lymphatic flow. Like other OMT procedures, it not only restores joint functions, but enhances positive well-being and full expression of a patient's life. In this technique, passive, smooth, rhythmic motion of the shoulder joint is done by the therapist to stretch contracted muscles, ligaments, and capsule (Babu And Putcha.,2022).
  Interventions: Procedure: spencer mscle energy technique

INTERVENTIONS:
Procedure: spencer mscle energy technique — The effectiveness of MET found in chronic capsulitis is due to its effect on relieving pain, ensuring ROM incretions, and developing functional activities due to the muscle contraction in a precise direction and in a monitored position over resistance to assist in improving joint range by advancing joint flexibility. This procedure is suggested for all joints with limited ROM (Butt & Tanveer, 2022).
  Other Names: spencer MET

SUMMARY:
Stiff shoulder is a painful and severely debilitating condition. The inflammatory contracture of the glenohumeral joint capsule in stiff shoulder restricts both active and passive range of motion, with loss of external rotation being especially characteristic of this condition (Dyer et al., 2023). Stiff shoulder is clinically described by the continuing onset of shoulder pain and advanced exacerbation of the shoulder joint leading to exertion in the higher extremity activity, significant disability, and functional restrictions. The most common symptom of a stiff shoulder is night pain, resulting in sleep impediment that leads to one-sided sleep on the uninfected shoulder (Mao et al., 2022).

Spencer technique is a standardized series of treatments with broad application to diagnose, treat and establish prognosis for restricted mobility in shoulder. It was developed by Spencer in 1961. It is a multistep technique that combines Spencer's positioning, sequencing, slow stretching of the shoulder complex within pain-free limits done by physical therapist while incorporating muscular energy with post-isometric contraction and relaxation (Babu And Putcha., 2022).

DETAILED DESCRIPTION:
thirty diabetic female patients with Stiff shoulder with ages 45-55 years:

Group A(study group) :

15 patients received Spencer Muscle Energy Technique along with postural exercise 3 times a week for 8 week.

Group B (control group) :

15 patients received Classical physiotherapy treatment includes Transcutaneous Electrical Nerve Stimulation (TENS) for 15 minutes hotpack on the painful area for 15 minutes along with postural exercise 3 times per week for 8 week.

ELIGIBILITY:
Inclusion Criteria:

* 1) Women's age between 45 to 55 years old 2)Suffering from stiff shoulder for 2-12 months (stage 1 and 2) confirmed by an orthopaedic specialist.

  3) Diagnosed as type 2 DM for at least 5 years. 4) No treatment other than analgesics

Exclusion Criteria:

* 1. cases of traumatic stiff shoulder. 2. Osteoporosis and malignance of shoulder region. 3. Neurological deficit affect shoulder function. 4. rheumatoid arthritis. 5. recurrent subluxation of shoulder. 6. cervical radiculopathy. 7. history of shoulder surgery. 8. vascular diseases.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
pain pressure threshold algometry | will be measured at baseline, and it will be measured after eight weeks
  Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold.
Visual Analogue Scale (VAS) | will be measured at baseline, and it will be measured after eight weeks
  was used to assess the severity of pain before and after treatment for both groups

SECONDARY OUTCOMES:
goniometer | will be measured at baseline, and it will be measured after eight weeks
  measures the available range of motion
SPADI (shoulder pain and disability index). | will be measured at baseline, and it will be measured after eight weeks
  It is a self-revealed measure created to assess shoulder pathological conditions

CONTACTS AND LOCATIONS:
Overall Officials: NESREEN GHAREEB, Vice Dean, Principal Investigator — Professor